CLINICAL TRIAL: NCT04864002
Title: TRIGGERING AND PROTECTIVE FACTORS OF BURNOUT IN MEDICAL RESIDENT PHYSICIANS IN A LOWER-MIDDLE-INCOME COUNTRY: A CROSS-SECTIONAL STUDY
Brief Title: TRIGGERING AND PROTECTIVE FACTORS OF BURNOUT IN MEDICAL RESIDENT
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Aysha Almas, Associate Professor, Aga Khan University
Other Study IDs: 5135_Med ERC-17
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Burnout, Professional
Keywords: Burnout; Residents; Medicine; Pakistan
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. only observational cross sectional study — No intervention done. only observational cross sectional study

SUMMARY:
Residents and interns are prone to emotional and physical exhaustion, also known as burnout. Burnout has not been studied much in physicians working in lower-middle income countries. We conducted this cross-sectional study at two institutes to determine the burden of burnout among internal medicine residents and to identify triggering and protective factors associated with burnout. An abbreviated version of the Maslach Burnout scale was used to measure burnout, and protective and triggering factors were recorded according to known factors.

ELIGIBILITY:
Inclusion Criteria:

- All residents of the internal medicine program at both institutes

Exclusion Criteria:

* Residents who were part of a flexible training program, working in shifts and those who had done less than six months of training were excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Internal Medicine residents working at two institutes
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Burnout | 1 year
  Burden of Burnout

SECONDARY OUTCOMES:
Triggering factors | 1 year
  Triggering factors for burnout
Protective factors | 1 year
  Protective factors for burnout

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No